CLINICAL TRIAL: NCT05083208
Title: A Single Arm, Multi-center, Phase Ib Clinical Trial of PI3Kδ Inhibitor Parsaclisib Combined With Chidamide for the Treatment of Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: PI3Kδ Inhibitor Parsaclisib Combined With Chidamide for the Treatment of Relapsed/Refractory Peripheral T-cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The clinical development of parsaclisib was stopped by it's manufacturer.
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYML06
Record Dates: First submitted 2021-09-18; First posted 2021-10-19 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: Relapsed/Refractory Peripheral T-cell Lymphoma; PI3Kδ inhibitor; Chidamide
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — parsaclisib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PI3Kδ inhibitor Parsaclisib plus Chidamide (Experimental): Parsaclisib is taken orally every day continuously, at approximately the same time every day, without food restriction, once a day.
  Chidamide is taken fixed 20mg twice a week with an interval of no less than 3 days, and taken 30 minutes after breakfast.
  Interventions: Drug: Parsaclisib; Drug: Chidamide

INTERVENTIONS:
Drug: Parsaclisib — Phase Ib: Parsaclisib is taken orally every day continuously, at approximately the same time every day, without food restriction, once a day. This stage follows the traditional "3+3" model. Parsaclisib is set at 10 mg/day, 15 mg/day, 20 mg/day 3 dose groups, starting from 10 mg/day, each group included 3 subjects. The final dose determined at this stage will be used in the Phase II study. Patients without progression or unacceptable toxicity after 8 weeks enter maintenance treatment.
  Maintain treatment: 2.5mg orally every day continuously, at approximately the same time every day, without food restriction, once a day until disease progression, death or unacceptable toxicity developments.
  Other Names: IBI376; PI3K inhibitor
Drug: Chidamide — Phase Ib: Chidamide is taken fixed 20mg twice a week with an interval of no less than 3 days, and taken 30 minutes after breakfast, until progression or intolerance.

SUMMARY:
This is a prospective single-arm, multicenter, phase Ib clinical trial of PI3Kδ inhibitor Parsaclisib combined with chidamide for the treatment of relapsed/refractory peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old (including 18 and 75)
2. Agreeing to sign the written informed consents
3. Diagnosed as peripheral T-cell lymphoma, including peripheral T-cell lymphoma, unspecified type, anaplastic large cell lymphoma (ALK negative or positive), angioimmunoblastic T-cell lymphoma, enteropathy Related T-cell lymphoma, hepatosplenic T-cell lymphoma, γ/δ T-cell lymphoma, NK/T-cell lymphoma, and other subtypes of PTCL that the investigator judges to be suitable for participating in this study
4. Received at least first-line anti-tumor therapy in the past, whether or not Chidamide has been used
5. Having at least one measurable lesions
6. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2
7. Life expectancy no less than 3 months
8. enough main organ function
9. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
10. Agreeing to follow the trail protocol requirements

Exclusion Criteria:

1. Types other than peripheral T-cell lymphoma listed in the enrollment criteria
2. Diagnosed as central nervous system lymphoma
3. Received palliative treatment for other malignant tumors in the past 2 years
4. Uncontrolled active infection
5. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
6. The non-hematological toxicity caused by the previous anti-tumor treatment has not recovered to ≤1 grade, and the hematological toxicity has not recovered to ≤2 grade
7. Patients with a history of mental illness
8. Those who are known to be allergic to the active ingredients or excipients of the drug parsaclisib and chidamide
9. Received PI3Kδ inhibitor treatment in the past
10. Received autologous hematopoietic or allogeneic hematopoietic stem cell transplantation within 3 months
11. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) >2
12. There are factors that affect the absorption of oral drugs
13. Pregnant or lactating women
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of Parsaclisib in Combination with Chidamide | Approximately 2 years
  This outcome measure will evaluate the safety and tolerability of parsaclisib when administered in combination with chidamide. Safety will be assessed by monitoring adverse events (AEs), dose-limiting toxicities (DLTs), and other clinically significant toxicities according to the Common Terminology Criteria for Adverse Events (CTCAE). Tolerability will be assessed based on the occurrence and severity of AEs during the trial, as well as the ability of patients to complete the treatment regimen without discontinuation due to adverse effects.
Recommended Phase 2 Dose (RP2D) of Parsaclisib in Combination with Chidamide | Approximately 2 years
  This outcome measure will determine the recommended Phase 2 dose (RP2D) of parsaclisib when combined with a fixed dose of 20 mg of chidamide administered twice weekly (BIW). The RP2D will be determined based on dose escalation, safety data, and the tolerability observed in the Phase Ib portion of the study. The RP2D will be the highest dose level at which no more than 33% of patients experience dose-limiting toxicities (DLTs) within the first treatment cycle.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, approximately 2 years
  The objective response rate will be calculated by dividing the number of patients who achieve CR or PR by the total number of patients in the study population.
Complete Response Rate (CRR) | Through study completion, approximately 2 years
  CRR will be reported as the proportion of patients who achieve CR among the total number of patients treated.
1-year progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment (each cycle is 28 days).
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first
1-year overall survival | from date of the first cycle of treatment to the date of death from any cause, assessed up to 2 years after last patient's enrollment (each cycle is 28 days).
  from date of first day of treatment to the date of death by any cause

OTHER OUTCOMES:
Correlation between baseline tumor gene mutation profile and clinical efficacy (CRR, PFS, OS) | Through study completion, approximately 2 years
  Baseline tumor tissue will be analyzed using a targeted next-generation sequencing (NGS) panel to determine the tumor gene mutation profile, including the presence of predefined somatic mutations. Clinical efficacy will be evaluated by complete response rate (CRR), progression-free survival (PFS), and overall survival (OS). The correlations between baseline tumor gene mutation profile and CRR, PFS, and OS will be explored using appropriate statistical methods (Fisher's Exact Test).
Correlation between tumor microenvironment characteristics assessed by single-cell sequencing, flow cytometry and clinical efficacy (CRR, PFS, OS) | Through study completion, approximately 2 years
  Tumor microenvironment characteristics will be assessed using single-cell sequencing and flow cytometry of tumor tissue and peripheral blood cells obtained at baseline (and, if available, at on-treatment time points). Parameters of interest include the composition and abundance of immune cell subsets (e.g., CD8+ T cells, regulatory T cells, NK cells, macrophage subpopulations) and their gene-expression signatures. These variables will be quantified as the proportion of each cell subset among total viable cells (%) or as gene-expression scores. Clinical efficacy will be evaluated by CRR, PFS, and OS as defined in the protocol.
  The correlations between tumor microenvironment features and clinical efficacy outcomes (CR and non-CR) will be explored using appropriate statistical methods (Independent t-test, Mann-Whitney U test, or ANOVA-two way).

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China